CLINICAL TRIAL: NCT04696978
Title: Metabonomics Characteristics and Predictive Value for Perioperative Neurocognitive Disorders After Deep Brain Stimulation Surgery for Parkinson's Disease
Brief Title: Study for Perioperative Neurocognitive Disorders After Deep Brain Stimulation Surgery for Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: wenbinlu (Other)
Responsible Party: Sponsor-Investigator, wenbinlu, Principal Investigator, Changhai Hospital
Organization: Changhai Hospital (Other)
Other Study IDs: PND-PD
Record Dates: First submitted 2020-12-23; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Neurocognitive Disorders
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — blood of patients is collected in normal patients and PND patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PND group: patients occur neurocognitive disorders according to scores in this group
- NO PND group: patients do not occur neurocognitive disorders according to scores in this group

SUMMARY:
Perioperative neurocognitive disorders(PND) is common to see in elderly patients. Although PND increases patient mortality as well as hospitalization time, apparent inflammatory factors, and related mechanisms are still unknown. Metabolites could reveal chemical fingerprints left behind by cellular processes, which in turn provide a new aspect to understand the biological process behind. we aim to found the metabolomics can aid the development of diagnostic markers of PND screening, early detection, and further, provide a basis for disease prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's patients undergoing elective deep brain stimulation
* Age ≥55 years
* ASA physical statusⅠ-Ⅲ
* Elementary school or above

Exclusion Criteria:

* patients with ASA physical status>III
* patients with systemic immune diseases, hematological diseases (hematological tumors or leukemia), patients after transplantation, malignant tumors
* patients with metabolic diseases such as diabetes, ketoacidosis, hyperosmolar syndrome, long-term hypoglycemia,gout
* patients who refused to join the study and lost to follow-up

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: we select Parkinson's patients undergoing elective DBS and observe who occur PND or not.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
the level of metabolomics in patients' blood sample | baseline
the level of metabolomics in patients' blood sample | 24 hours after operation
the level of metabolomics in patients' blood sample | 72 hours after operation

SECONDARY OUTCOMES:
CAM-ICU score | baseline
CAM-ICU score | 24 hours after operation
CAM-ICU score | 72 hours after operation
CAM-ICU score | 1 month after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, Shanghai Municipality, China